CLINICAL TRIAL: NCT02459535
Title: Immediate and Long-term Induction of Incretin Release by Artificial Sweeteners 1
Acronym: ILIAS-1
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: German Institute of Human Nutrition (Other)
Collaborators: Ludwig-Maximilians - University of Munich (Other)
Responsible Party: Principal Investigator, Prof. Dr. med. Andreas F. H. Pfeiffer, Director, Department of Clinical Nutrition, German Institute of Human Nutrition
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: ILIAS-1
Record Dates: First submitted 2015-03-23; First posted 2015-06-02 (Estimated); Last update posted 2020-06-24 (Actual); Status verified 2020-06

CONDITIONS: Pre-diabetes; Diabetes
Keywords: incretin release
MeSH Terms: conditions — Glucose Intolerance; Diabetes Mellitus

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (7):
- Glucose only (Active Comparator): oral ingestion of 54 g Glucose in 300 ml water at t=0 in fasted state; blood samples over 120 mins
  Interventions: Other: oral stimulation glucose
- Glucose + Saccharin (Active Comparator): oral ingestion of 54 g Glucose + 0,112 g Saccharin in 300 ml water at t=0 in fasted state; blood samples over 120 mins
  Interventions: Other: oral stimulation glucose; Other: oral stimulation saccharin
- Saccharin only (Active Comparator): oral ingestion of 0,112 g Saccharin in 300 ml water at t=0 in fasted state; blood samples over 120 mins
  Interventions: Other: oral stimulation saccharin
- Glucose + Aspartame (Active Comparator): oral ingestion of 54 g Glucose 0,197 g Aspartame in 300 ml water at t=0 in fasted state; blood samples over 120 mins
  Interventions: Other: oral stimulation glucose; Other: oral stimulation aspartame
- Aspartame only (Active Comparator): oral ingestion of 0,197 g Aspartame in 300 ml water at t=0 in fasted state; blood samples over 120 mins
  Interventions: Other: oral stimulation aspartame
- Glucose + Sucralose (Active Comparator): oral ingestion of 54 g Glucose + 0,088 g Sucralose in 300 ml water at t=0 in fasted state; blood samples over 120 mins
  Interventions: Other: oral stimulation glucose; Other: oral stimulation sucralose
- Sucralose only (Active Comparator): oral ingestion of 0,088 g Sucralose in 300 ml water at t=0 in fasted state; blood samples over 120 mins
  Interventions: Other: oral stimulation sucralose

INTERVENTIONS:
Other: oral stimulation glucose — oral stimulation with glucose, AS or glucose+AS in fasted state, blood samples from fasted state up to 120 min post-ingestion
  Arms: Glucose + Aspartame; Glucose + Saccharin; Glucose + Sucralose; Glucose only
Other: oral stimulation saccharin
  Arms: Glucose + Saccharin; Saccharin only
Other: oral stimulation aspartame
  Arms: Aspartame only; Glucose + Aspartame
Other: oral stimulation sucralose
  Arms: Glucose + Sucralose; Sucralose only

SUMMARY:
Epidemiological data suggest, that not only sugar-based, but also artificially sweetened soft drinks may play a role in the development of diabetes.

Recent studies in animals and humans have shown, that artificial sweeteners (AS) influence metabolic responses after glucose ingestion, possibly alter the intestinal microbiome and even modulate incretin release.

However, it is unclear, if these findings are valid for all kinds of AS, as they are chemically different. Furthermore, data on human subjects are sparse and controversial.

The investigators will therefore conduct 7 consecutive single oral stimulations with glucose or AS alone or a combination. Three different AS will be tested.

DETAILED DESCRIPTION:
Epidemiological data suggest, that not only sugar-based, but also artificially sweetened soft drinks may play a role in the development of diabetes.

Recent studies in animals and humans have shown, that artificial sweeteners (AS) influence metabolic responses after glucose ingestion, possibly alter the intestinal microbiome and even modulate incretin release.

However, it is unclear, if these findings are valid for all kinds of AS, as they are chemically different. Up to now, no single study has ever compared metabolic responses to different AS in the same subjects. Furthermore, data on human subjects are sparse and controversial. This is partially explained by different methodical approaches such as intragastral/intraduodenal application of AS, rather than conventional oral consumption.

The investigators will therefore conduct 7 consecutive single oral stimulations with glucose or AS alone or a combination. Three different AS will be tested: saccharin, aspartame and sucralose.

ELIGIBILITY:
Inclusion Criteria:

* healthy

Exclusion Criteria:

* metabolic disorders such as diabetes, hypothyroidism, corticoid therapy, heart or lung disease

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 14 (Actual)
Dates: Start 2015-03 (Actual); Primary Completion 2017-06 (Actual); Study Completion 2019-07 (Actual)

PRIMARY OUTCOMES:
change in GIP release | 120 mins
  comparison between all seven interventions
change in GLP-1 release | 120 mins
  comparison between all seven interventions
change in GLP-2 release | 120 mins
  comparison between all seven interventions
change in PYY release | 120 mins
  comparison between all seven interventions
change in insulin release | 120 mins
  comparison between all seven interventions
change in combined blood levels of glucose and insulin, expressed in calculated indices for insulin secretion | 120 mins
  comparison between all seven interventions
change in combined blood levels of glucose and insulin, expressed in calculated indices for insulin sensitivity | 120 mins
  comparison between all seven interventions

CONTACTS AND LOCATIONS:
Locations (1):
- German Institut for Human Nutrition; Department for Clinical Nutrition, Bergholz-Rehbrücke, Brandenburg, Germany